CLINICAL TRIAL: NCT00243724
Title: An Open-Label, Parallel-Group, Multi-Centre Study to Determine the Effect of Treatment With Esomeprazole for Six Months on Histological Markers of Esophageal Epithelial Acid-Related Disease in Patients With Upper GI Symptoms.
Brief Title: HEARD (Long Term) Study - Histology of the Esophagus in Acid-Related Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00078
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Gastroesophageal Reflux; Heartburn; Dyspepsia
Keywords: immunohistochemical; erosive esophagitis; Acid reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Dyspepsia | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
Determine if different levels of acid-suppression with esomeprazole for 6 months on chosen histological markers of esophageal epithelial acid-related disease in patients with upper GI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 18 years or older
* history of upper GI symptoms

Exclusion Criteria:

* Peptic ulcer disease
* upper gastrointestinal surgery
* malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline after 6 months in the level of ki-67 expression and histological markers of esophageal epithelial acid-related disease after acid-suppressive therapy with esomeprazole

SECONDARY OUTCOMES:
Changes in immunohistochemical markers of esophageal epithelial acid-related disease after 6 months treatment with different levels of acid suppression with esomeprazole

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Canada Medical Director, MD, Study Director — AstraZeneca
Locations (10):
- Canada (10):
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Guelph, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, North York, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec